## Application form for non-AMG/non-MPG studies

## (in addition, a separate study protocol must be submitted)

(See also "explanations of the application for non-AMG/non-MPG studies)

| 1 | Applicant: Name, Address, Tel./Fax-No.: | |
|---|---|---|
| | Tepsanti ramo, radioos, rom ak-non | Dr. med. Monika Empl Neurology Consultant Department of Neurology Department of Neurology Ludwig-Maximilians University Munich University Hospital Munich-Großhadern Marchioninistraße 15 D- 81377 Munich Tel.: +49 89-4400-73906 E-mail: monika.empl@med.uni- muenchen.de |
| | | UnivProf. Dr. med. Andreas Straube Senior Physician Department of Neurology Ludwig-Maximilians University Munich University Hospital Munich-Großhadern Marchioninistraße 15 D- 81377 Munich Telephone: +49 89-4400-73900 E-Mail: Andreas.Straube@med.uni- muenchen.de UnivProf. Dr. Angelika C. Wagner Pedagogic Psychology Department of educational science Research Group Introvision, University of Hamburg Bogenallee 11 D - 20144 Hamburg Telephone: +49 40-42838-7990 E-Mail: Angelika.Wagner@uni- |
| | | hamburg.de |
| 2 | Title of the research project: | Introvision in migraines and headaches-<br>IntroMig |
| 3 | Training data and research experience: | See enclosed application, page 2f |
| 4 | Monocentric or multicenter study: | |
| | In multicenter studies: | Monocentric study ⊗ multicenter study O |
| | Head of the clinical trial of other test centres, central evaluation point Votes of other ECs | - n.a |

| 5 | Declaration that the principles of the Helsinki Declaration are taken into account in their current version. | I/we declare that the principles of the Helsinki Declaration are taken into account in the current version |
|---|---|---|
| | | Munich, 22.10.2015 |
| | | (Dr. med. Monika Empl,<br>On behalf of all applicants) |
| 6 | Study-related burdens: | |
| | a) Radiation exposure | Yes O<br>No ⊗ |
| | <u>If yes:</u> | I/we declare that prior to the study the approval of the BFS is obtained. |
| | b) Diagnostic investigations | Yes O<br>No ⊗ |
| | c) Blood/Tissue Collection | Yes O<br>No ⊗ |
| 7 | Wissenschaftliche Angaben zum Forschungsvorhaben: | See enclosed application, page 3ff |
| 7.1 | Study Objective | See enclosed application, page 5f |
| 7.2 | Study Design | With control group Yes ⊗ No O |
| | | With healthy volunteers Yes O No ⊗ |
| _ | Case number estimation and evaluation acept | Yes ⊗ Mrs. Dr. Hoster, Institute for Biometry and Epidemiology (IBE), LMU See enclosed application, page 7f |

| | No O Please explain |
|---|---|
| 7.4 Statistical advice by | Mrs Dr. Hoster, IBE, LMU Munich |
| 7.5 Study duration | Expected Start Date: 01.12.2015 |
| | Expected End: 31.12.2016 |
| 8 Discussion of ethical-legal issues | See enclosed application, page 8 |
| 8.1. Discussion of the disadvantages, risks, burdens and potential benefits of the study | |
| 8.2. Inclusion of persons not able to consent | Provided O Not provided |
| <u>If provided:</u> | Indication of reasons |
| 8.3. Research on minors | Provided O Not provided ⊗ |
| <u>If provided:</u> | Indication of reasons |
| 9 Data protection | Irreversible anonymised use of samples/data (without reference to persons) |
| If pseudonymised use | pseudonymised use of samples/ persons) ⊗ Encryption) |
| | Information on how the encryption code is formed, who has access to the encryption code, reasons for decryption and how long the data/samples be kept |
| | See enclosed application, page 8f |
| 10 Insurance: | Declaration that an insurance policy is / was completed O |
| | Why insurance is not necessary ⊗ |
| | See enclosed application, page 9 |
| | A road insurance has been completed |

| | Yes O<br>No ⊗ |
|---|---|
| 11 Financing: A) Financing of the research project B) rewarding doctors/patients/volunteers | See enclosed application, page 9 |
| 12 Expenditure compensation for the EC: | The costs of expenditure compensation are taken over |
| | Application for reduction of expenditure compensation (explanation to attach) ⊗ |
| | Billing address (if different from the address of the applicant): |
| Date, Signature | 22.10.2015 |